CLINICAL TRIAL: NCT06189703
Title: tRNS Treatment for ADHD Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Innosphere (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TRNS-CLIN-003
Record Dates: First submitted 2023-12-19; First posted 2024-01-03 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: ADHD
Keywords: Pediatric
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, sham-controlled between groups
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study is double-blind, meaning participants, parents/legal guardians/caregivers, the investigator and all study personnel are blinded. Participants will be randomized in a 1:1 allocation ratio to receive active (Group A) or sham (Group B) tRNS. Randomization will be stratified by age, gender, and baseline ADHD-RS score. Three staff members with no contact with participants will generate balanced random samples throughout the course of the study, using Smith's randomization algorithm based on the variance minimization procedure, and program the respective device to discharge sham/active stimulation according to each participant's allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Group A: Treatment Arm (Active Comparator): The same device placement will be used for sham as in the active arm.
  Interventions: Device: tRNS
- Group B: Sham-Control Arm (Sham Comparator): The same device placement will be used for sham as in the active arm.
  Interventions: Device: tRNS

INTERVENTIONS:
Device: tRNS — transcranial random noise stimulation applied to the right IFG and the left DLPFC
  Other Names: Novostim 2

SUMMARY:
A randomized, sham-controlled, double-blind clinical trial to examine the safety and effectiveness of tRNS on unmedicated pediatric patients (7-12 years) with ADHD. Subjects will undergo either tRNS or sham treatment for 10 days during a two-week period in a home-simulated environment. Each treatment session is 20 minutes, during which their attention will be maintained using a software game.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Age between 7-12 years old at the time of enrollment
2. Estimated Full Scale IQ ≥ 85 based on WASI-II (Two-subtests Form) NOTE: Results of an equivalent and validated IQ test that were performed in the previous 12 months from the date of enrollment are acceptable. The Investigator must ensure that no significant head injuries, particularly significant head trauma, occurred in this period from the previous test to the enrollment.
3. Score above the standard clinical cut-off score for ADHD symptoms on the ADHD DSM-5 scales
4. Meet criteria for ADHD according to DSM-5, using the "gold standard" procedure as described by the American Academy of Pediatrics, which includes a semi-structured interview of the subject and parent(s)/legal guardian(s)
5. Moderate to severe ADHD as defined as having a minimum score of 12 on either the inattention subscale or the and hyperactivity-impulsivity subscale of the baseline ADHD Rating Scale (ADHD-RS), and a Clinical Global Impression-Severity (CGI-S) score at baseline of greater than 4
6. Parent(s)/legal guardian(s) fluent in English, able to complete ADHD-RS scale and attend all study visits
7. Has not taken any medication with central nervous system effects, including prescription medications for ADHD, within 7 days of enrollment, as determined by the investigator based on the subject's medical history from the parent(s)/legal guardian(s) and, as applicable, medical and pharmacy records

EXCLUSION CRITERIA:

1. Has a history of any medical or psychiatric disorder, disease, condition, injury, symptoms or circumstance that, in the opinion of the principal investigator, may: (1) reduce the subject's ability to fulfill the study requirements as per protocol; or (2) adversely impact the integrity of the data or the validity of the study results
2. Primary DSM-5 axis-1 disorder other than ADHD, which consists of one or more of severe ODD, bipolar psychosis, major depressive disorder, severe oppositional defiant disorder that would pose adherence challenges by the investigator
3. Substance abuse, that, in the opinion of the investigator, may: (1) reduce the participant's ability to fulfill the study requirements as per protocol; or (2) adversely impact the integrity of the data or the validity of the study results
4. Impaired functioning to a degree that requires immediate initiation of ADHD medication in the opinion of the Investigator
5. Known hypersensitivity to Polyamide or Elastomer
6. Any suicide risk as assessed with the Columbia-Suicide Severity Rating Scale (Pediatric (≤11 years) Quick Screen)
7. If female, began menstruation, based on a self- or parent(s)/legal guardian(s)-report
8. Any other condition, which would make the participant unsuitable to participate in this study as determined by the Investigator
9. Inability to provide informed consent and assent (participant and parent(s)/legal guardian(s))

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 146 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in ADHD symptom severity during treatment | Baseline to End of Treatment (Week 2)
  Change in ADHD symptom severity, measured by total score of parent-reported ADHD-RS questionnaire from baseline to End of Treatment (Week 2) compared to sham control.
Incidence of adverse events | Baseline to Week 10
  Incidence of adverse events (AEs), including serious adverse events (SAEs) related to Novostim 2 treatment

SECONDARY OUTCOMES:
Change in ADHD symptom severity post-treatment | Baseline to Follow-up 1 (Week 4) and to Follow-up 2 (Week 10)
  Change in ADHD-RS from baseline to follow-up (Week 4 and Week 10) compared to sham control
Change in ADHD-RS subscales | Baseline to End of Treatment (Week 2), Follow-up 1 (Week 4) and Follow-up 2 (Week 10)
  Change in ADHD-RS subscales (either inattention or hyperactivity-impulsivity subscales) from baseline to end of treatment and follow-up (Week 4 and Week 10) compared to sham control
GCI-I score | Baseline to End of Treatment (Week 2), Follow-up 1 (Week 4) and Follow-up 2 (Week 10)
  CGI-I score at end of treatment and follow-up (Week 4 and Week 10) compared to sham control

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Boston Children's Hospital, Boston, Massachusetts
  - Mayo Clinic Hospital, Methodist Campus, Rochester, Minnesota
  - Baylor College of Medicine Department of Psychiatry & Behavioral Sciences, Houston, Texas
  - UTHealth Houston, Houston, Texas
- Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No